CLINICAL TRIAL: NCT06462339
Title: Investigation of the Effects of Online Pilates Training on Cognitive Functions and Dual-Task Performance in Multiple Sclerosis Patients
Brief Title: The Effect of Online Pilates on Cognitive Function and Dual-Task Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Kader Eldemir, Principal Investigator, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-Cognition-Onlinepilates
Record Dates: First submitted 2024-05-24; First posted 2024-06-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cognitive Function; Dual-task; Pilates; Telerehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Two groups as exercise group and control group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates training via telerehabilitation (Experimental): The intervention group will be received online pilates training three times a week for 6 weeks.
  Interventions: Behavioral: Experimental: Intervention Group
- Waitlist (No Intervention): The control group will be a wait-list group without any additional specific treatment.

INTERVENTIONS:
Behavioral: Experimental: Intervention Group — The group that will receive pilates training via telerehabilitation
  Arms: Pilates training via telerehabilitation

SUMMARY:
Multiple sclerosis (MS) is a chronic, inflammatory, degenerative disease of the central nervous system, causing demyelination and axonal damage. MS typically begins with attacks resulting from demyelination of axons, eventually evolving into a neurodegenerative disease associated with neurotrophic support deficiency and neuronal loss. Depending on the location and degeneration, various neurological disorders and symptoms such as walking and balance problems, fatigue, sensory loss, and cognitive impairments are observed in MS patients. Cognitive impairments in MS are associated with lesion count, localization, axonal loss, and brain atrophy, affecting approximately 50-60% of patients. Patients exhibit impairments in verbal fluency, visual-spatial memory, processing speed, executive functions, and episodic memory. Cognitive impairments also lead to a decrease in dual-task performance, referred to as the ability to perform two tasks simultaneously, in MS patients. Cognitive problems and impaired dual-task performance negatively impact various aspects of daily life, including social participation and employment status, thus reducing their quality of life.

Clinical-based exercise interventions are frequently utilized and effective in improving cognitive functions and dual-task performance in MS. Pilates is a commonly used exercise modality in clinical practice. Pilates is a core stability-based exercise method involving endurance, flexibility, movement, posture, and respiratory control. Previous studies have indicated that clinical Pilates improves cognitive functions. On the other hand, telerehabilitation approaches, the use of which has increased rapidly due to technological developments in recent times, enable the delivery of rehabilitation services to patients in distant places by using communication technologies. For this purpose, it is highly valuable to implement Pilates, which consists of core stability exercise content, through telerehabilitation. While there are studies on clinical-based Pilates interventions, no study has investigated the efficacy of one-on-one online Pilates exercises on cognitive functions and dual-task performance in an online platform. Therefore, this study aims to investigate the effects of online Pilates on cognitive functions and dual-task performance in patients with MS.

DETAILED DESCRIPTION:
This study is a randomized controlled study. The patients will be randomly divided into two groups exercise and control. Pilates exercises consisting of 3 days a week for 6 weeks will be given to the exercise group.

The control group will be a wait-list group without any additional specific treatment.

All assessments will be done before and after the 6-week intervention program or waiting period. The demographic characteristics of the participants initially will be taken and the Expanded Disability Status Scale score of those of MS will be recorded. As the outcome measures, cognitive functions and dual-task performance will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Voluntarily participate in research to accept
* Having a diagnosis of "Multiple Sclerosis" by a specialist physician
* Relapse free in the last 3 mounts
* An Expanded Disability Status Scale (EDSS) score: 0-5

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, hearing, and perception problems that may affect the results of the research
* Having a cardiovascular, pulmonary or hormonal disorder that would prevent exercise
* Having an accompanying neurological disorder other than MS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-11-12 (Actual)

PRIMARY OUTCOMES:
Mini-Mental test-Baseline | Assessment will be conducted before the intervention
  Mini Mental Test (MMT) consists of eleven items grouped under five main headings: orientation, recording memory, attention and calculation, recall and language, and is evaluated out of a total score of 30. Accordingly, getting 24 points and above is considered normal.
Mini-Mental test-Post intervention | Assessment will be conducted immediately after the intervention
  Mini Mental Test (MMT) consists of eleven items grouped under five main headings: orientation, recording memory, attention and calculation, recall and language, and is evaluated out of a total score of 30. Accordingly, getting 24 points and above is considered normal.
Montreal Cognitive Assessment-Baseline | Assessment will be conducted before the intervention
  The Montreal Cognitive Assessment (MoCA) was developed as a rapid screening test for mild cognitive impairment. MoCA evaluates different cognitive functions. These; attention and concentration, executive functions, memory, language, visual structuring skills, abstract thinking, calculation and orientation. The highest total score that can be obtained from the test is 30. Higher scores mean a better outcome.
Montreal Cognitive Assessment-Post intervention | Assessment will be conducted immediately after the intervention
  The Montreal Cognitive Assessment (MoCA) was developed as a rapid screening test for mild cognitive impairment. MoCA evaluates different cognitive functions. These; attention and concentration, executive functions, memory, language, visual structuring skills, abstract thinking, calculation and orientation. The highest total score that can be obtained from the test is 30. Higher scores mean a better outcome.
Trail Making Test-Baseline | Assessment will be conducted before the intervention
  Trail Making Test (TMT) is used to evaluate individuals' executive functions, task-sequence switching ability, attention, visual scanning speed, visual-motor perception, planning, organization, abstract thinking and reaction limitation. The test consists of 2 parts: A and B. In part A, the individual is asked to combine numbers from 1 to 25 and the completion time is recorded. In part B, the individual completes the sequence corresponding to a number and a letter respectively, and the completion time is recorded.
Trail Making Test-Post intervention | Assessment will be conducted immediately after the intervention
  Trail Making Test (TMT) is used to evaluate individuals' executive functions, task-sequence switching ability, attention, visual scanning speed, visual-motor perception, planning, organization, abstract thinking and reaction limitation. The test consists of 2 parts: A and B. In part A, the individual is asked to combine numbers from 1 to 25 and the completion time is recorded. In part B, the individual completes the sequence corresponding to a number and a letter respectively, and the completion time is recorded.
Stroop Test-Baseline | Assessment will be conducted before the intervention
  Stroop Test, one of the neuropsychological tests, is used to evaluate selective attention, information processing speed and cognitive flexibility. The test consists of three parts. The first section contains words written in black (e.g. 'blue'), the second section contains colors, and the last section contains words written in different colors (e.g. the word blue written in red ink). The participant is expected to fulfill the tasks in these three sections respectively. While keeping time for each part, the participant must read the words correctly at first, say the colors in the next part, and say the color in which the word is written in the last part. In the test, reading time, number of errors made and number of spontaneous corrections are recorded.
Stroop Test-Post intervention | Assessment will be conducted immediately after the intervention
  Stroop Test, one of the neuropsychological tests, is used to evaluate selective attention, information processing speed and cognitive flexibility. The test consists of three parts. The first section contains words written in black (e.g. 'blue'), the second section contains colors, and the last section contains words written in different colors (e.g. the word blue written in red ink). The participant is expected to fulfill the tasks in these three sections respectively. While keeping time for each part, the participant must read the words correctly at first, say the colors in the next part, and say the color in which the word is written in the last part. In the test, reading time, number of errors made and number of spontaneous corrections are recorded.
Functional mobility-baseline | Assessment will be conducted before the intervention
  Timed up and go test measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again.
Dual task performance in functional mobility, Cognitive additional task (arithmetic)-baseline | Assessment will be conducted before the intervention
  Timed up and go test measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again.
  Cognitive additional task (arithmetic): Individuals will be asked to perform tasks by counting backward from 3 to 3 from 100.
Dual task performance in functional mobility, Cognitive additional task (verbal)-baseline | Assessment will be conducted before the intervention
  Timed up and go test measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again.
  Cognitive additional task (verbal): Individuals will be asked to fulfill their duties by producing name.
functional mobility-post intervention | Assessment will be conducted immediately after the intervention
  Timed up and go test measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again.
Dual task performance in functional mobility, Cognitive additional task (arithmetic)-post intervention | Assessment will be conducted immediately after the intervention
  Timed up and go test measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again.
  Cognitive additional task (arithmetic): Individuals will be asked to perform tasks by counting backward from 3 to 3 from 100.
Dual task performance in functional mobility, Cognitive additional task (verbal)-post intervention | Assessment will be conducted immediately after the intervention
  Timed up and go test measures the time taken in seconds to arise from a standard chair, walk 3 m, turn through 180 degrees, walk back, and sit down again.
  Cognitive additional task (verbal): Individuals will be asked to fulfill their duties by producing name.
balance-baseline | Assessment will be conducted before the intervention
  The posturography (Biodex Balance System-BioSwayTM) will be used to assess postural stability.
balance, Cognitive additional task (arithmetic)-baseline | Assessment will be conducted before the intervention
  The posturography (Biodex Balance System-BioSwayTM) will be used to assess postural stability.
  Cognitive additional task (arithmetic)
Dual task performance in balance, Cognitive additional task (verbal)-baseline | Assessment will be conducted before the intervention
  The posturography (Biodex Balance System-BioSwayTM) will be used to assess postural stability.
  Cognitive additional task (verbal)
Dual task performance in balance,Cognitive additional task (arithmetic)-post intervention | Assessment will be conducted immediately after the intervention
  The posturography (Biodex Balance System-BioSwayTM) will be used to assess postural stability.
  Cognitive additional task (arithmetic)
balance-post intervention | Assessment will be conducted immediately after the intervention
  The posturography (Biodex Balance System-BioSwayTM) will be used to assess postural stability.
Dual task performance in balance,Cognitive additional task (arithmetic) -post intervention | Assessment will be conducted immediately after the intervention
  The posturography (Biodex Balance System-BioSwayTM) will be used to assess postural stability.
  Cognitive additional task (arithmetic)
Dual task performance in balance,Cognitive additional task (verbal) -post intervention | Assessment will be conducted immediately after the intervention
  The posturography (Biodex Balance System-BioSwayTM) will be used to assess postural stability.
  Cognitive additional task (verbal)
gait-baseline | Assessment will be conducted before the intervention
  Wearable system (G-Walk) will be used to assess gait parameters.
Dual task performance in gait, Cognitive additional task (arithmetic)-baseline | Assessment will be conducted before the intervention
  Wearable system (G-Walk) will be used to assess gait parameters. Cognitive additional task (arithmetic)
Dual task performance in gait, Cognitive additional task (verbal)-baseline | Assessment will be conducted before the intervention
  Wearable system (G-Walk) will be used to assess gait parameters. Cognitive additional task (verbal)
gait-post intervention | Assessment will be conducted immediately after the intervention
  Wearable system (G-Walk) will be used to assess gait parameters.
Dual task performance in gait, Cognitive additional task (arithmetic)-post intervention | Assessment will be conducted immediately after the intervention
  Wearable system (G-Walk) will be used to assess gait parameters. Cognitive additional task (arithmetic)
Dual task performance in gait, Cognitive additional task (verbal)-post intervention | Assessment will be conducted immediately after the intervention
  Wearable system (G-Walk) will be used to assess gait parameters. Cognitive additional task (verbal)

CONTACTS AND LOCATIONS:
Overall Officials: Kader Eldemir, PT, MSc., Study Chair — Ordu University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analysis of all data are made, all results will be shared

REFERENCES:
- [Background] Abasiyanik Z, Ertekin O, Kahraman T, Yigit P, Ozakbas S. The effects of Clinical Pilates training on walking, balance, fall risk, respiratory, and cognitive functions in persons with multiple sclerosis: A randomized controlled trial. Explore (NY). 2020 Jan-Feb;16(1):12-20. doi: 10.1016/j.explore.2019.07.010. Epub 2019 Jul 17. PMID 31377306
- [Background] Ozkul C, Guclu-Gunduz A, Eldemir K, Apaydin Y, Yazici G, Irkec C. Combined exercise training improves cognitive functions in multiple sclerosis patients with cognitive impairment: A single-blinded randomized controlled trial. Mult Scler Relat Disord. 2020 Oct;45:102419. doi: 10.1016/j.msard.2020.102419. Epub 2020 Jul 23. PMID 32736216
- [Derived] Eldemir K, Eldemir S, Ozkul C, Irkec C, Guclu-Gunduz A. The effects of online pilates training on cognitive functions and dual task performance in people with multiple sclerosis: A randomized controlled study. Mult Scler Relat Disord. 2025 May;97:106393. doi: 10.1016/j.msard.2025.106393. Epub 2025 Mar 17. PMID 40120159